CLINICAL TRIAL: NCT06797401
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Trial Evaluating the Efficacy and Safety of RBD5044 in Patients With Mixed Dyslipidemia
Brief Title: Phase 2 Trial Evaluating the Efficacy and Safety of RBD5044 in Patients With Mixed Dyslipidemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ribocure Pharmaceuticals AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC02T001; 2023-510369-92 (EudraCT Number)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Dyslipidemias
Keywords: Mixed dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (participant, care provider, investigator, outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose group (Experimental): Participants will receive RBD5044 or placebo as subcutaneous injections at Day 1 and Day 84.
  Interventions: Drug: RBD5044; Drug: Placebo
- Medium dose group (Experimental): Participants will receive RBD5044 or placebo as subcutaneous injections at Day 1 and Day 84.
  Interventions: Drug: RBD5044; Drug: Placebo
- High dose group (Experimental): Participants will receive RBD5044 or placebo as subcutaneous injections at Day 1 and Day 84.
  Interventions: Drug: RBD5044; Drug: Placebo

INTERVENTIONS:
Drug: RBD5044 — RBD5044, active drug.
Drug: Placebo — Placebo that is identical in appearance and volume to the doses of active IMP.

SUMMARY:
The goal of this clinical trial is to learn if drug RBD5044 works to treat mixed dyslipidemia in adults. It will also learn about the safety of drug RBD5044. The main questions it aims to answer are:

Does drug RBD5044 reduce the triglyceride levels? What medical problems may participants experience when taking drug RBD5044? Researchers will compare drug RBD5044 to a placebo to see if drug RBD5044 works to treat mixed dyslipidemia.

Participants will:

Receive RBD5044 or placebo twice during the trial (Day 1 and Day 84). Visit the clinic 11 times during 12 months (visit every 4-8 weeks) for checkups and tests.

DETAILED DESCRIPTION:
This is a multicentre, randomised, double-blinded, placebo-controlled, parallel-group phase 2 clinical trial to evaluate the efficacy and safety of RBD5044 subcutaneous injections in participants with mixed dyslipidemia.

There will be 3 different dose level groups of RBD5044 or placebo: low dose (n=40), medium dose (n=40) or high dose (n=40). Within each of the 3 dose cohorts, participants will be randomly assigned in a 3:1 ratio to either active (RBD5044) treatment or to placebo treatment. All trial groups will be dosed in parallel.

All participants will be dosed at their trial site and undergo blood sampling and examinations at pre-defined timepoints.

Participants will be followed-up for 48 weeks from the first day of IMP/placebo administration. Primary endpoint evaluation will take place in week 16. End of trial is in week 48.

ELIGIBILITY:
Inclusion Criteria:

* Willing to comply with protocol required visit schedule and visit requirements and provide written informed consent.
* Male or female participants, aged 18 to 80 years inclusive.
* Fasting TG level of ≥ 150 mg/dL (≥ 1.69 mmol/L) and <499 mg/dL (5.61 mmol/L).
* Fasting levels at screening of non-HDL-C ≥ 100 mg/dL (2.59 mmol/L), or low-density lipoprotein cholesterol (LDL-C) ≥70 mg/dL (1.8 mmol/L) after at least 4 weeks of stable diet and stable optimal statin therapy (+ or - ezetimibe) if indicated.
* Body mass index between 18 and 40 kg/m2.

Exclusion Criteria:

* Any uncontrolled or serious disease, or any medical or surgical condition, that may interfere with participation in the clinical trial and/or put the participant at significant risk (according to the investigator's judgment) if he/she participates in the clinical trial.
* Uncontrolled hypertension (blood pressure >160/100 mmHg at screening). (If untreated, participant may be re-screened once hypertension is treated and controlled).
* Active or history of serious mental illness or psychiatric disorder, including but not limited to schizophrenia, bipolar disorder, or severe depression, which require current pharmacological intervention. Participants with a history of severe depression who are no longer on medication.
* Any of the following laboratory values at screening:

Hepatic: ALT or AST >2× ULN at screening, eGFR <30 mL/min/1.73 m2 (using the Modification of Diet in Renal Disease [MDRD] equation) at Screening, HbA1c >9.0% (or >75 mmol/mol International Federation of Clinical Chemistry [IFCC] units) at screening.

* Patients with a diagnosis of HBV, HCV or HIV at screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in triglyceride (TG) levels at week 16 | From baseline until end week 16
  Percent change from baseline in TG levels at week 16.

SECONDARY OUTCOMES:
Frequency, intensity and seriousness of the AEs during the trial | Each visit from baseline to week 48 (end of trial)
  Number and percentage of participants with AEs. All reported AE terms will be coded using Medical Dictionary for Drug Regulatory Affairs (MedDRA).
Change from baseline in triglyceride (TG) levels at different time points | week 4, 8, 12, 20, 24, 32, 40 and 48
  Percent change from baseline in TG levels at different time points
Change from baseline in ApoC-III levels at different time points | week 4, 8, 12, 20, 24, 32, 40 and 48
  Percent change from baseline in ApoC-III levels at different time points
Plasma concentrations of RBD5044 | In conjunction of administration of the IMP
Change from baseline in lipid parameters levels at different time points | week 4, 8, 12, 16, 20, 24, 32, 40 and 48
  Percent change from baseline in TC, LDL-C, HDL-C, non-HDL-C, TRL-C, ApoB, ApoA1, Lp (a) levels at different time points

CONTACTS AND LOCATIONS:
Overall Officials: Sara Svedlund, MD, PhD, Principal Investigator — Ribocure Clinic/Ribocure Pharmaceuticals AB; David Erlinge, MD, PhD, Principal Investigator — Lunds Universitetssjukhus; Emil Hagström, MD, PhD, Principal Investigator — Akademiska Sjukhuset Uppsala
Locations (3):
- Sweden (3):
  - Lunds Universitetssjukhus, Lund
  - Ribocure Clinic/Ribocure Pharmaceuticals AB, Mölndal
  - Akademiska Sjukhuset Uppsala, Uppsala

IPD SHARING:
Plan to Share IPD: No